CLINICAL TRIAL: NCT05824598
Title: OsteopaThic, logopedIc and Psychological Assessment To Improve Outcome in pAtieNts undergoIng Cardiac Surgery: a Randomized Clinical Trial (TITANIC Trial)
Brief Title: Multifunctional Approach in Cardiac Surgery
Acronym: TITANIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06_08/02/2023
Record Dates: First submitted 2023-03-13; First posted 2023-04-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-03

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: cardiac surgery; cardiac rehabilitation; swallowing disorders; post-surgical pain; psychological counseling; osteopathic manipulative treatment
MeSH Terms: conditions — Deglutition Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Monocentric, single blind with parallel arm design. Standard descriptive analysis and linear and logistic regression models will be performed.
  To correct any imbalances between the 2 groups due to the low sample size, an analysis adjusted for the main confounders listed below is planned: age, gender, previous cognitive impairment, previous presence of anxiety and depression beyond the clinically acceptable threshold.
  Sample size estimation was performed using G*Power v3.1 software. The sample size was calculated separately for the two outcomes of interest that will make up the composite score: reduction in pain assessed using the Numerical Rating Scale (NRS) and reduction in anxiety and depression assessed using the Hospital Anxiety and Depression Scale (HADS).
  It was then decided to conservatively adopt the higher number of the two estimates.
Who Masked: Outcomes Assessor
Masking Description: The pain scores will be assessed by a psychologist blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The cases (active treatment) will be treated with an approach that includes osteopathic treatment for pain control (by the Osteopath Bruno Bordoni), systematic swallowing screening (Speech Therapist, Leone Stilo), psychological counseling (Psychologist, Eleonora Volpato, Giulia Novembre ). The duration of treatment will be that of hospitalization, on average about 3 weeks. The osteopathic treatment will last 5 sessions, while the counseling will have one session at the admission and one at the discharge and up to two sessions a week (variable according to individual needs); the swallowing screening will have one session at the admission and one at discharge and about two-three sessions a week (variable according to individual needs).
  Interventions: Behavioral: Multifunctional rehabilitation treatment
- Controls (No Intervention): Controls will follow good clinical practice (in this case systematic screening from a swallowing point of view will not be applied, nor will osteopathic treatment and systematic psychological counseling be considered).

INTERVENTIONS:
Behavioral: Multifunctional rehabilitation treatment — multidisciplinary approach with (OMT, psychological counseling, and therapists dedicated to swallowing disorders)
  Arms: Treatment

SUMMARY:
Postoperative pain and swallowing disorders are complex, multifactorial phenomenon that frequently occur after cardiac surgery. Preoperative anxiety and the interaction between sex and other sociocultural factors may predict greater sensitivity to postoperative pain, whereas the epidemiology and course of swallowing disorders has not been systematically investigated, along with the interaction between dysphagia, post-operative pain and emotional stress. Cardiac rehabilitation is a multifunctional intervention which may address all these functional domains, improving patients' prognosis.

The aim of the present study is to demonstrate the superiority of a multifunctional approach (OMT, systematic swallowing screening and specific treatment according to good clinical practice associated with psychological counseling) compared to local clinical practice in the management of pain and swallowing disorders.

DETAILED DESCRIPTION:
The TITANIC trial will provide evidence on whether a multifunctional intervention systematically implemented in the cardiac rehabilitation setting will improve the clinical course and prognosis of patients with recent cardiac surgery.

The design is a randomized clinical trial with parallel group design. Patients aged over 18 undergoing elective cardiac surgery and admitted to IRCCS Fondazione Don Gnocchi, Santa Maria Nascente, Milan, for cardiac rehabilitation will be randomized to standard post-acute treatments (cardiovascular training, monitoring and logopedic treatment only in case of swallowing dysfunction) compared with an experimental approach which consists of osteopathic manipulative treatment (OMT) treatments, swallowing screen protocol, psychological assessment and counseling.

This study may help in the identification of a new diagnostic-therapeutic pathway in cardiac surgery patients that allows a reduction in the use of analgesics and anti-inflammatories and increases the early detection of swallowing disorders. Furthermore, by allowing an integrated assessment of emotional needs, it can have a positive effect in reducing the need for post-operative clinical visits and assessments in the medium to long term, improving the patients' quality of life.

ELIGIBILITY:
Inclusion Criteria (all the following must be satisfied):

* patients with recent cardiac surgery (within one month)
* without swallowing disorders already identified before discharge
* with the presence of chest pain (NRS>2).

Exclusion Criteria:

* patients who are unable to sign informed consent.
* patients with already known psychological/psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pain release through the Brief Pain Inventory | Through study completion, an average of 4 weeks
  To verify the effectiveness of the multifunctional rehabilitation approach in reducing pain assessed by the Brief Pain Inventory: likert scale with maximum pain intensity equal to 7-10.
Anxiety and depression control through the Hospital Anxiety and Depression Scale | Through study completion, an average of 4 weeks
  To verify the effectiveness of the multifunctional rehabilitation approach in reducing anxiety and depression assessed by the Hospital Anxiety and Depression Scale (HADS), with maximum anxiety and depression equal to 15-21 points.

SECONDARY OUTCOMES:
To assess functional swallowing disorders post-cardiac surgery (Mealtime Assessment Scale) | Through study completion, an average of 4 weeks
  Epidemiological framework of the cardiac surgery population, in terms of presence/absence of swallowing disorders. MAS: points 0-36, with higher scores defining the worst outcome.
Anti-inflammatory drugs use (numbers of pills used) | Through study completion, an average of 4 weeks
  Monitoring the use of anti-inflammatory drugs
LOS | Through study completion, an average of 4 weeks
  Length of stay
Number of participants with persistent inflammatory status | Through study completion, an average of 4 weeks
  The persistent inflammatory status will be described in terms of fever and PCR> 5 in at least two successive measurements 8 days apart)
Adherence to treatment | Through study completion, an average of 4 weeks
  Monitoring of adherence to treatment using the 4-item Morisky, Green, and Levine Adherence Scale. With a sum of scores of 8, from 6 to <8 or <6, patients can be classified as having high, medium or low adherence to therapy, respectively.
Quality of life improvement through the EuroQol Visual Analogue Scale (EuroQoL-VAS) questionnaire | Through study completion, an average of 4 weeks
  Consisting of two parts. The first explores 5 areas of interest: mobility, personal hygiene, social activities, pain and anxiety/depression. Each individual area has, in turn, three levels of severity (no problem, problem of some size, problem of extreme seriousness). The second section consists of a 20 cm visual analog scale (VAS) on which the patient indicates the best (score=0) or worst (score=100) possible state of health.
Cognitive impairment | Through study completion, an average of 4 weeks
  Monitoring of cognitive abilities through the administration of the Montreal Cognitive Assessment Test (MOCA) scale, with a score more than 17,54 in the normal range. A raw and then corrected score: - less than 15.5 suggests the presence of a cognitive impairment;
  - between 15.5 and 17.54 assumes a borderline performance; - a score above 17.54 would show functioning within the normal range.
Quality of life improvement through the Short Form-12 (SF-12) questionnaire | Through study completion, an average of 4 weeks
  Scores can be reported as Z-scores (difference from the population mean, measured in standard deviations). The population mean is 50 points. The population standard deviation is 10 points. Thus, each 10-point increase above or below 50 is one standard deviation from the mean.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Gnocchi, ONLUS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No